CLINICAL TRIAL: NCT04135040
Title: Assessment of the Protein Quality of Cereal Grains in School-aged Children
Brief Title: Lysine Metabolic Availability in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H17-00452
Record Dates: First submitted 2018-06-04; First posted 2019-10-22 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Children
Keywords: IAAO; Lysine; Children; Cereal Grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lysine metabolic availability (Experimental): Lysine metabolism from pure amino acids and cereal foods in children.
  Interventions: Dietary Supplement: L-Amino Acid

INTERVENTIONS:
Dietary Supplement: L-Amino Acid — 8 different lysine intakes (L-Amino Acid and food) will be tested for 8 hours each.

SUMMARY:
This study will evaluate how much of the essential amino acid lysine school-aged children are using for protein synthesis when consuming different cereal grains. Six healthy children between 6-10y will be recruited. They will be given cooked white rice, corn, oats, black beans, and milk. Using a minimally invasive technique, the amount of lysine that is available from cereal grain products will be determined. With the results from this research project accurate diet recommendations will be developed for children consuming cereal-based diets.

DETAILED DESCRIPTION:
Purpose The purpose of this research project is to implement the minimally invasive Indicator Amino Acid Oxidation (IAAO) method in healthy school-aged children to measure the metabolic availability of the essential amino acid lysine obtained from commonly consumed cereal grains and their breakfast counterparts. Additionally, the difference in metabolic availability through complementation of breakfast cereals with milk will be assessed.

Hypothesis The use of the IAAO method will yield a higher lysine metabolic availability for those cereal grains that have the least amount of fibre in the food matrix. Combining the consumption of cereals with milk will increase the metabolic availability of lysine.

Justification Cereal grains and their derived products are the most commonly consumed food group around the world. From traditional foods such as steamed rice, corn tortillas, and wheat bread to relatively modern products like ready-to-eat breakfast cereals. Up to 80% of the energy intake in developing countries comes from this food group. Given that they are considered as a low protein quality food source, a considerable amount of the world's population could potentially be at risk of lysine deficiency. Especially, children living in underdeveloped countries where complementation with other food sources, such as legumes, dairy, or other animal products, is not an available option. Since lysine is the limiting amino acid in cereals, this study is of great importance not only for its nutritional value, but also for its social and economic impact.

Current lysine recommendations for school-aged children are based on factorial calculations performed on results of adult male studies. To develop the Lysine EAR (Estimated Average Requirement) for growing children, these studies use adult lysine maintenance requirements multiplied by estimated rates of protein deposition and the efficiency of this deposition. Additionally, these studies do not measure lysine's bioavailability, which will vary depending on the food sources and the processing techniques used to preserve them. With these limitations in mind, the IAAO method has the capacity to accurately measure amino acid metabolic availability in different populations groups, such as healthy and malnourished children. Metabolic availability refers to the amount of absorbed amino acids that are used for protein synthesis. It takes into account all amino acid losses from digestion, absorption, metabolic utilization, and endogenous losses.

Previously, this method was used to determine lysine metabolic availability of rice in healthy adults. This is the only study of this nature done for any human food source. Currently, there is no information available regarding lysine's metabolic availability from corn, wheat, milk and any breakfast cereal. Previously the IAAO method has successfully been implemented in healthy Canadian and Indian children to measure lysine requirements. Additionally, lysine requirement studies has been preformed in moderately undernourished Indian children with parasitic intestinal infections. The study conclusions were that, undernourished children require around 20% more lysine than their healthy counterparts. In these cases it is not only important to know the lysine content of a food source, but also it's metabolic availability, to develop accurate interventions that will have a better chance to meet children's daily requirements.

Given that childhood is a critical period for optimal growth and development, a comprehensive study of lysine's metabolic availability in commonly consumed cereal grains is needed to develop adequate interventions and recommendations, targeted to prevent stunting and other signs of malnourishment in at risk populations around the world.

Objective The general objective of this research project is to assess the degree in which cereal food sources can meet lysine amino acid requirements in healthy school-aged children.

The specific objective us to:

- Determine the metabolic availability of lysine from rice, corn, oats, black beans and milk using the IAAO method in healthy school-aged children.

Research Design This is a repeated measures study design involving 1 pre-study visit and 8 study visits approximately one week apart from each other.

ELIGIBILITY:
Inclusion Criteria:

* Healthy school-aged children between the ages of 6-10y.
* Normal weight.
* Normal eating habits.

Exclusion Criteria:

* Children under 6 years old, or over 10 years old.
* Children who are currently ill (fever, cold, vomiting or diarrhea).
* Children outside normal weight parameters (3rd - 85th percentiles for weight).
* Children with claustrophobia.
* Children currently or recently taking medication or antibiotics.
* Children with food allergies.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
13 CO2 production | 8 hours (1 study day)
  Breath samples will be collected during the study day, to measure the rate of oxidation of tracer phenylalanine in the expired breath.

SECONDARY OUTCOMES:
Urinary lysine | 8 hours, 2 samples at the beginning and end of the study day.
  Urine will be collected during the study day to measure urinary excretion of lysine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other researchers

REFERENCES:
- [Derived] Caballero K, Mandal R, Pratap-Singh A, Kitts DD, Ball RO, Pencharz PB, Courtney-Martin G, Elango R. Lysine Bioavailability in School-Age Children Consuming Rice Is Reduced by Starch Retrogradation. J Nutr. 2020 Dec 10;150(12):3208-3215. doi: 10.1093/jn/nxaa276. PMID 33025006